CLINICAL TRIAL: NCT01349686
Title: Fluid Oral Intake vs. Fasting During Labour: A Randomized, Controlled Trial.
Brief Title: Effect of Fluid Oral Intake During Labour
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator of Research, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MHST2011-03
Record Dates: First submitted 2011-05-05; First posted 2011-05-06 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Labor
Keywords: Food; Fluids; Labor
MeSH Terms: interventions — Diet; Angptl4 protein, mouse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral intake of fluids (Experimental): Intake of oral fluids during labour.
  Interventions: Procedure: Diet
- Fasting (Placebo Comparator): No intake of oral fluids during labour.
  Interventions: Procedure: Fasting

INTERVENTIONS:
Procedure: Diet — Oral intake of fluids during labour, from admission (dose: two cups of 8 ounces each of clear tea with little sugar).
  Arms: Oral intake of fluids
Procedure: Fasting — No intake of fluids during labour.
  Arms: Fasting

SUMMARY:
Fasting during labour is a usual conduct in many hospitals around the world (due to the theorical risk of bronchoaspiration). There is little evidence supporting this conclusion. Besides, there are several studies that suggest that food intake during labour can be associated with shorter labours and a lower cesarean rate. The aim of the investigators study is to show if the oral intake of fluids during labour can reduce the first stage of labour with minimum risk to the patient.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age > 37 weeks.
* Cervical dilation < 5 cms.

Exclusion Criteria:

* Maternal pathologies (diabetes, heart disease, preeclampsia)
* Breech presentation or any other condition that is an indication of cesarean section.
* Premature rupture of membranes.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2011-09; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Duration of labour (measured in minutes from admission to delivery) | Two months

SECONDARY OUTCOMES:
Number of cesarean sections due to prolonged second stage of labour (measured in number of cases). | Two months
Number of cases of bronchoaspiration. | Two months

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Espinosa, Resident, Principal Investigator — Saint Thomas Hospital, Panama; Osvaldo Reyes, Doctor, Principal Investigator — Saint Thomas Hospital, Panama
Locations (1):
- Saint Thomas Hospital, Panama City, Provincia de Panamá, Panama